CLINICAL TRIAL: NCT01114061
Title: Evaluation of the Effects of Heating the Vicinity of the Insulin Delivery Site by the InsuPatch Device During Daily Life
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Insuline Medical Ltd. (Industry)
Responsible Party: Ingabriel bitton, Insuline Medical LTD.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HT4813
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes
Keywords: diabetes; postprandial glucose level; insulin pharmacodynamics; Insulin Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- InsuPatch (Experimental): The arm with the treatment: using the insupatch device to heat the insulin infusion site.
  Interventions: Device: Insupatch

INTERVENTIONS:
Device: Insupatch — Applying heat to the infusion site using the insupatch device

SUMMARY:
The aim of this study is to test the performance of the InsuPatch device in daily life. The primary target of the study is to evaluate safety aspect of daily device use. Additional aspects to be evaluated in the study are: the effect of the device on post prandial glucose level.

DETAILED DESCRIPTION:
Despite the recent years advance in rapid acting insulin analogues early postprandial hyperglycemia and late post prandial hypoglycemia are still common in insulin treated diabetic patients. It appears that even with these rapid acting insulins there is still a significant delay time and variability in the delay time between the changes in blood glucose levels following the meals and the absorption kinetics of insulin injected subcutaneously. Past studies using regular human insulin have demonstrated that using local stimulation at the injection site can dramatically improve regular insulin kinetics. The assumption was that local stimulation induces local increase in blood perfusion which improves insulin absorption from the injection site.

Following the above Insulin has developed the InsuPatch device. The intended use of the InsuPatch device is to improve insulin delivery into the blood when the insulin is infused using an insulin-infusion pump by controlled heating of the area surrounding the point of infusion.

The InsuPatch device consists of two components:

I) InsuPatch single-use, flat, heating pad with electrical wire which is attached by adhesive to the bottom of the Medtronic MiniMed Quick-set® infusion set. The user attaches the device to the infusion set prior to insertion of the infusion set catheter.

II) The InsuPatch case is used as a case for the Medtronic MiniMed Paradigm insulin infusion pump. The InsuPatch case contains an electronic unit and batteries.

The effect of the device on the pharmacokinetics (PK) and pharmacodynamics (PD) of the injected insulin were tested in Euglycemic clamp and meal tolerance test (MTT) studies. The effect of the device on insulin PK was evaluated by comparing insulin concentration in the meal MTT study with and without operation of the device. The effect of the device on insulin PD was evaluated using Euglycemic clamp protocol with and without operation of the device. The effect of the device on postprandial glucose excursions was tested by comparing the post meal glucose levels with and without operation of the device.

The main results of the study were:

1. An increase of 49% in the available insulin in the blood during the first 30 minutes post injection and 37% in during the first hour post injection (PK).
2. A reduction of 25% in the average glucose level during post-meal first two hours (PD).
3. A reduction of 43% in the time to peak action of insulin (PD).

The aim of this study is to test the performance of the InsuPatch device in daily life. The primary target of the study is to evaluate safety aspect of daily device use. Additional aspects to be evaluated in the study are: the effect of the device on post prandial glucose level.

ELIGIBILITY:
Inclusion Criteria:

1. Participant age between 18- 65 years old (including = 18 years and =65 years)
2. BMI: 18-35 kg/m2
3. Insulin dependent diabetes under insulin pumps.
4. Use of short-acting insulin analogues
5. Subjects agreeing to use the InsuPatch device.
6. 6% ≤ HbA1c ≤ 9.5%
7. Agree to sign consent form.
8. Subject is willing to do at least 4 blood glucose recordings per day
9. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
10. Willing to comply with all specified follow-up evaluations

Exclusion Criteria:

1. Pregnancy
2. Breast feeding women.
3. Alcohol addiction
4. Had CABG (Coronary Artery Bypass Graft), Post MI (Myocardial Infarction) or had active Ischemic heart disease in the last 3 months prior to the study date
5. Had CVA (cardiovascular accident) or TIA (transient ischemic accident) in the last 12 months prior to the study
6. Suffer from Hypertension (blood pressure > 140/90) .
7. Low blood hemoglobin concentration <9 g/dL for female and <11g/dL for male.
8. Known gastro- or enteroparesis
9. Abnormal kidney and/ or liver function tests. (Creatinine >1.5 mg/dL, liver test> 2 times the upper limit of the normal range).
10. Severe hypoglycemic events requiring glucagon injection or glucose infusion within the last six months prior to study inclusion
11. Hypoglycaemia unawareness
12. Diabetic ketoacidosis (severe, with hospitalization) within the last six months prior to study inclusion
13. Psychological incompetence
14. Signs of drug abuse
15. Any other clinical condition or history, that seems to be relevant to the principle investigator to disqualify the participant.
16. Not willing to sign the inform consent form.
17. Subjects with diminished skin integrity, Excessive fibrosis, lipo-hypertrophy or eczema at infusion sites
18. Subjects with heat sensitivity
19. Subjects involved in or planed to participate in other studies.
20. Any subject whom the primary researcher consider not suited to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
show no increase in hypoglycemia events when the InsuPatch device is used compared to the number of hypoglycemia events when the InsuPatch device is not used. | three month with the device and three months without the device
  Show that the hypoglycemia rate is not increased when the InsuPatch device is used